CLINICAL TRIAL: NCT00233311
Title: Assessment of the Postprandial Effects of a Fast-food on Inflammatory Markers
Brief Title: Fast Food Study: Assessment of the Effects of Fast-Food on Inflammatory Markers
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: AG0052
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Heart Diseases; Diabetes; Obesity
Keywords: high fat diet; inflammation; inflammatory markers; C-reactive protein; Aging
MeSH Terms: conditions — Heart Diseases; Diabetes Mellitus; Obesity; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Whole Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to determine whether eating a fast food meal (high in saturated fat) will result in greater increases in inflammatory markers than eating a meal with low levels of saturated fat and higher levels of mono-unsaturated fat. This study is a first step in learning about how dietary fat intake can directly impact risk factors for heart disease, diabetes and obesity.

DETAILED DESCRIPTION:
At the first visit, each potential participant will undergo the screening examination, including laboratory tests. An electrocardiogram (ECG) is performed at baseline to exclude participants with evidence of myocardial infarction. Each participant will complete a Food Intake Record to assess typical dietary patterns. Cognitive status will be assessed with the Mini-Mental Status Exam. The potential participant must acknowledge his or her willingness to consume the two test meals designed for the study.

During visits 2 and 3, the participant will undergo the Oral Glucose Tolerance Test. The Fast Food and Healthy Meals will be administered during Visits 4,5,6 & 7. After fasting for at least 8 hours, the participant will have an intravenous (IV) line placed in an arm vein. Twenty minutes will be allotted for participants to complete each experimental meal (either the fast food or healthy meal). At the end of the 20 minutes, blood will be collected through an intravenous port over an eight-hour time period. Baseline blood samples will also be collected prior to each meal. The two mixed meals will be: 1) a fast-food meal equivalent to the Big Mac Meal with French fries and milkshake; 2) a meal with the same fat distribution as the fast-food meal with fats derived from mono-unsaturated fat sources. A registered dietitian will prepare both of the meals. To prevent any carry-over effects from previous meals, participants will be asked to fast overnight with their last meal being a light dinner no later 12 hours before scheduled testing. In addition, participants will be asked to avoid high fat, high calorie meals during the course of the study. Participants will be given specific dietary guidelines to follow during the course of the study and in the four days preceding the OGTT at visit 2. They will be asked to complete a diet diary so that their adherence to the dietary recommendations can be monitored. All participants will be asked to continue with their normal exercise routine with the exception that no exercise is to be done in the 24 hours prior to each testing session. During the OGTT and the testing sessions for the two meals, an ECG will be continuously recorded using a Holter monitor.

The primary study hypotheses are:

* Administration of the different meals (different nutrient compositions) will cause differential increases in the circulating levels of inflammatory markers. Specifically, the fast-food meal (high in saturated fat) will cause a greater increase in circulating inflammatory markers, specifically C-reactive protein (CRP), than the oral glucose or the mono-unsaturated fat meal. Also, this difference in inflammatory response will not be explained by parallel changes in circulating lipid levels.
* The inflammatory response within an individual to the standard oral glucose tolerance test (OGTT) and to each meal is reproducible over a 48-hour period.

The secondary hypothesis is:

* Changes in the serum level of glucose and insulin following a standard oral glucose tolerance test will predict changes in circulating levels of inflammatory markers after both meals

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women between the ages of 50 and 65
* Body mass index (BMI) less than or equal to 30 kg/m2
* Waist circumference less than or equal to 40 inches for men and 35 inches for women (measured at natural waist just above the navel)
* CRP (C-reactive protein) level less than 3mg/L
* Report no difficulties or need for help in performing self care or instrumental activities of daily living
* Able to walk for at least 10 minutes without needing to stop or without symptom onset
* No substantial cognitive impairment based on mental status screening tests (score <24 on Mini-Mental Status Exam)
* No history of a cardiovascular event over the last three months (including angina, myocardial infarction, coronary artery bypass graft surgery (CABG), congestive heart failure, cerebro-vascular diseases), cancer, diabetes mellitus, neurological disease, thyroid disease, birth defect, kidney or liver disease, gastrointestinal (G.I.) diseases (including gallbladder disease), musculoskeletal disorder (if they cause pathological weakness and/or chronic pain), or important sensory deficits.

Exclusion Criteria:

* Systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than or equal to 95 mmHg with or without treatment
* ECG shows evidence of myocardial infarction
* Abnormal laboratory tests
* Abnormal liver function
* Shortness of breath while performing normal activities of daily living, such as walking or climbing stairs
* Use of any hormones (i.e. estrogen, testosterone)
* Absolute need for long-term treatment with anti-inflammatories, aspirin (>100 mg per day per physician orders), statins, antibiotics, corticosteroids, immunosuppressors, H2 blockers and pain medications. Non-steroid anti-inflammatory use is allowed, but should be stopped three days before the study)
* Use of herbal supplements are not permitted during the study (Multivitamin is permitted, but other vitamin supplementation are not permitted during the study.)
* Any medication/drug that acts on lipid metabolism (i.e. Xenical)
* Any severe psychiatric condition
* Any infections requiring use of antibiotics within the past 3 months
* Current use of tobacco products
* Alcoholic intake > 30 grams while on this study is not permitted (no more than 2 beers per day or more than one glass of wine or cocktail daily)
* Intense physical activity over the past year (>6 metabolic equivalents [METs], at least 1 hour per week)
* Allergies to nuts
* Loss or gain of greater than or equal to 4 pounds in the past 6 months
* Any condition that may preclude informed consent
* Recent blood donation (past 3 months)

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General Public
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2004-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Ferrucci, MD, PhD, Principal Investigator — MedStar Research Institute, NIA/Astra Unit, National Institute on Aging
Locations (1):
- NIA Clinical Research Unit at Harbor Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Bender R, Jockel KH, Trautner C, Spraul M, Berger M. Effect of age on excess mortality in obesity. JAMA. 1999 Apr 28;281(16):1498-504. doi: 10.1001/jama.281.16.1498. PMID 10227319
- [Background] Carroll MF, Schade DS. Timing of antioxidant vitamin ingestion alters postprandial proatherogenic serum markers. Circulation. 2003 Jul 8;108(1):24-31. doi: 10.1161/01.CIR.0000074221.68903.77. Epub 2003 Jun 23. PMID 12821556
- [Background] Cohn JS, McNamara JR, Cohn SD, Ordovas JM, Schaefer EJ. Postprandial plasma lipoprotein changes in human subjects of different ages. J Lipid Res. 1988 Apr;29(4):469-79. PMID 3392464
- [Background] de Bruin TW, Brouwer CB, van Linde-Sibenius Trip M, Jansen H, Erkelens DW. Different postprandial metabolism of olive oil and soybean oil: a possible mechanism of the high-density lipoprotein conserving effect of olive oil. Am J Clin Nutr. 1993 Oct;58(4):477-83. doi: 10.1093/ajcn/58.4.477. PMID 8379502
- [Background] Festa A, D'Agostino R Jr, Howard G, Mykkanen L, Tracy RP, Haffner SM. Chronic subclinical inflammation as part of the insulin resistance syndrome: the Insulin Resistance Atherosclerosis Study (IRAS). Circulation. 2000 Jul 4;102(1):42-7. doi: 10.1161/01.cir.102.1.42. PMID 10880413